CLINICAL TRIAL: NCT04771585
Title: Quantification of Exhaled Particles to Identify Airborne Transmission Risks of SARS-Co-V-2
Brief Title: Quantification of Exhaled Particles to Identify Airborne Transmission Risks of COVID-19
Acronym: QUELLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 20-14 QUELLE
Record Dates: First submitted 2021-01-26; First posted 2021-02-25 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Healthy
Keywords: Aerosols; Exhaled particles; Face mask

STUDY DESIGN:
Intervention Model Description: In part A of the study, aerosol emission of subjects will be characterized. From this population, the 10 highest-emitting subjects will enter part B of the study to investigate the effect of face masks on aerosol emission down to the submicron range.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Part A (No Intervention): Aerosol number and size spectrum characterization of 30 subjects, stratified by age groups, including 10 professional singers. Subjects will be examined twice within 14 days to assess reproducibility of aerosol emission.
- Study Part B (Experimental): From the 30 subjects of Part A, the 10 highest-emitting subjects will be assessed a third time, wearing four different classes of face masks consecutively with increasing aerosol filtering capacity.
  Interventions: Other: Community Mask; Other: Surgical Mask; Other: FFP2 respirator; Other: FFP3 respirator

INTERVENTIONS:
Other: Community Mask — Fabric mask, no medical device
  Arms: Study Part B
Other: Surgical Mask — Medical face mask (personal protective equipment), CE-certified
  Arms: Study Part B
Other: FFP2 respirator — Filtering Face Piece with no less than 94% filtering capacity, CE-certified
  Arms: Study Part B
Other: FFP3 respirator — Filtering Face Piece with no less than 99% filtering capacity, CE-certified
  Arms: Study Part B

SUMMARY:
In this study, the aerosols emitted during various respiratory activities will be quantified in healthy subjects. The differences in aerosol size spectrum and number during tidal breathing, speaking, coughing and singing will be assessed. Subjects with an endogenously high aerosol emission will repeat the respiratory activities wearing face masks with varying particle filter capacity to investigate the aerosol emission reduction.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give written informed consent.
2. Healthy male and female subjects, aged 18-80 years.
3. Body mass index between 18 and 35 kg/m2.
4. FEV1 ≥ 80% predicted.

Exclusion Criteria:

1. Any clinically relevant abnormal findings in physical examination or lung function at screening visit, which, in the opinion of the investigator, may either put the subject at risk because of participation in the study or may influence the results of the study, or the subject's ability to participate in the study.
2. Risk of non-compliance with study procedures.
3. Suspected inability to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study.
4. History of an acute respiratory infection with symptoms such as cough, rhinitis, sore throat, hoarseness or fever, within four weeks prior to the informed consent visit. In case of acute respiratory infection during study participation, the visit may be rescheduled within the allowed time window. Subjects must be asymptomatic for at least 3 days. Re-screening is allowed should the time window be exceeded.
5. History of lung disease including but not confined to COPD, asthma or pulmonary fibrosis.
6. History of latex allergy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
To compare the emitted small particle fraction between various respiratory activities. | Day 1, Day 2 to 14
  Change of particle number per time unit between tidal breathing and various respiratory activities.
To assess the influence of different face masks on the emitted small particle fraction of various respiratory activities. | After completion of Study part A (approximately 3 months)
  Change of particle number per time unit between tidal breathing and selected respiratory activities for community masks, surgical masks, FFP2 and FFP3 respirators in high-emitting subjects.

SECONDARY OUTCOMES:
To assess the emitted particle size distribution of various respiratory activities. | Day 1, Day 2 to 14
  Compare changes of emitted particle size spectrum as quantity per size range during tidal breathing and selected respiratory activities.
To assess the reproducibility of exhaled particle quantification. | Day 2 to 14
  Compare results for particle number per time unit and particle size spectrum from visit 1 and 2.
To assess the influence of different face masks on the emitted particle size distribution of various respiratory activities. | After completion of Study part A (approximately 3 months)
  Compare changes of emitted particle size spectrum as quantity per size range during tidal breathing and selected respiratory activities for community masks, surgical masks, FFP2 and FFP3 respirators in high-emitting subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Fraunhofer ITEM, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schwarz K, Struss N, Banari L, Hohlfeld JM. Quantifying Exhaled Particles in Healthy Humans During Various Respiratory Activities Under Realistic Conditions. J Aerosol Med Pulm Drug Deliv. 2024 Apr;37(2):51-63. doi: 10.1089/jamp.2022.0076. Epub 2024 Jan 29. PMID 38285475